CLINICAL TRIAL: NCT06231745
Title: The GRK2 Inhibitor Paroxetine as a Novel Adjunct to Conventional Therapy in Rheumatoid Arthritis Patients.
Brief Title: Paroxetine Safety and Efficacy in Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Teaching assisstant, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 314879
Record Dates: First submitted 2024-01-20; First posted 2024-01-30 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Paroxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): group one (control group): 50 patients will receive the conventional DMARDs therapy (methotrexate 7.5 mg IM once weekly) plus placebo tablets
  Interventions: Drug: Methotrexate
- Comparative group (Active Comparator): 50 patients will receive the conventional DMARDs therapy (methotrexate 7.5 mg IM once weekly) plus 20 mg paroxetine daily
  Interventions: Drug: Methotrexate; Drug: Paroxetine

INTERVENTIONS:
Drug: Methotrexate — Methotrexate (MTX) is an anti-metabolite most commonly used in chemotherapy and immunosuppressant in auto-immune diseases. This activity describes the indications, action, and contraindications for Methotrexate as a valuable agent in treating a wide variety of diseases.
Drug: Paroxetine — Paroxetine is a type of antidepressant known as a selective serotonin reuptake inhibitor (SSRI). It's often used to treat depression, and sometimes obsessive compulsive disorder (OCD), panic attacks, anxiety or post-traumatic stress disorder (PTSD).
  Arms: Comparative group

SUMMARY:
Rheumatoid arthritis (RA) is a systemic chronic auto-inflammatory disorder which imposes a remarkable burden of morbidity and mortality on global health. The complex interaction between genetics, environment, and immunological response contribute to RA pathogenesis. Current treatment comprises conventional disease-modifying anti-rheumatic drugs (DMARDs) followed by biological DMARDs, if necessary, to achieve low disease activity or remission. Therapeutics used in RA had limitations in tolerability, access, and response duration and magnitude. Consequently, implementation of safe adjunctive treatment for RA is urgently needed to boost the therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* Aged 23-57 years fulfilling 2010 American College of Rheumatology - European League against Rheumatism (ACR-EULAR) classification criteria for RA (12) and had active inflammatory RA with no limit in disease duration.
* Patients received MTX, nonsteroidal anti-inflammatory drugs, selective cyclooxygenase-2 inhibitors, acetaminophen, and low dose of oral corticosteroids will be allowed to enroll the trial
* Intravenous, intra-articular or intramuscular corticosteroids; intra-articular hyaluronate sodium; biological DMARDs; and other DMARDs will not be permitted less than 4 weeks before the first dose of paroxetine.

Exclusion Criteria:

* patients refusing to give informed consent, diabetes, congestive heart failure, previous adverse reaction to paroxetine, oral prednisolone greater than 10 mg/day, receiving biological DMARDs, severe anemia, active infection, pregnancy or lactation, and clinically significant renal or hepatic disease.

Ages: 23 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy end point will be the change in the 28-joints disease activity score (DAS28). | 3 months
  A DAS28 value of greater than 5.1 indicates high disease activity. The values of 3.2 < DAS28 ≤ 5.1 and DAS28 ≤ 3.2 are indicative of moderate and low disease activities, respectively. If DAS28 value is less than 2.6, the patients may be considered to be in remission phase

CONTACTS AND LOCATIONS:
Locations (1):
- Mostafa Bahaa, Damietta, New Damietta, Egypt

REFERENCES:
- [Derived] Aldossary KM, Abdallah MS, Mosalam EM, Kamal N, Saif DS, Elsayed SA, Afifi N, Zakaraia HG, Khrieba MO, Bahaa MM. Efficacy of Paroxetine as an Adjuvant Therapy in Rheumatoid Arthritis Patients: A Randomized Controlled Study. Drug Des Devel Ther. 2025 Dec 30;19:11925-11939. doi: 10.2147/DDDT.S572677. eCollection 2025. PMID 41488752